CLINICAL TRIAL: NCT00526552
Title: RAPID (Evaluating the Efficacy of RosuvAstatin for Korean Dyslipidemia PatIents With Diabetes in Real World Practice)
Brief Title: Crestor RAPID (The Efficacy of RosuvAstatin for Korean Dyslipidemia PatIents With Diabetes)
Acronym: RAPID
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-CKR-CRE-2007/3
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Dyslipidemia; Diabetes
Keywords: dyslipidemia; rosuvastatin; diabetes; cholesterol; Naturalistic; Observational
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the efficacy of rosuvastatin in Korean dyslipidemia patients with diabetes

ELIGIBILITY:
Inclusion Criteria:

* Hyperlipidemia patients who are prescribed with rosuvastatin 10mg, based on clinical grounds and fulfil the following criteria

  1. Over 18 years of age
  2. Diagnosed with DM based on fasting or post-load glucose data and/or clinical assessment by the clinician

Exclusion Criteria:

1. Patients already taking other hyperlipidemic agents
2. Patients who do not fulfil the indication criteria for statin therapy
3. Patients who do not have baseline and/or follow-up lipid data to verify the efficacy data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic Mellitus patients with hypercholesteromia in Korean tertiary care centers
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2007-06; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyunah Caroline Choi, Study Director — AstraZeneca Korea
Locations (3):
- South Korea (3):
  - Research Site, Seoul, Jongro-gu
  - Research Site, Seoul, Kangnam-gu
  - Research Site, Seoul, Songpa-gu